CLINICAL TRIAL: NCT04905719
Title: Reliability of Point-of-Care Ultrasound Examination in Primary Care Performed by a General Practitioner
Brief Title: Point-of-Care Ultrasound in Primary Care
Acronym: POCUS iGP 1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Emergency Medical Service of the Central Bohemian Region, Czech Republic (Other)
Collaborators: The Society of General Practice, J. E. Purkyne Czech Medical Association (Unknown); Institute for Postgraduate Medical Education, Czech republic (Unknown)
Responsible Party: Principal Investigator, Roman Skulec, Principal Investigator, Emergency Medical Service of the Central Bohemian Region, Czech Republic
Other Study IDs: POCUSiGP01
Record Dates: First submitted 2021-05-24; First posted 2021-05-28 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with dyspnea: Patients who visit a general practitioner for dyspnea will undergo a Point-of-Care ultrasound examination of the lungs to identify the presence or the absence of A-profile, B-profile and pleural effusion.
  Interventions: Diagnostic Test: Ultrasound
- Patients with abdominal pain: Patients who visit a general practitioner for abdominal pain in the right upper quadrant will undergo abdominal Point-of-Care ultrasound examination to identify cholecystolithiasis.
  Interventions: Diagnostic Test: Ultrasound
- Patients with suspected deep vein thrombosis: Patients who visit a general practitioner for pain and / or swelling of the lower extremity will undergo compression ultrasound testing to identify proximal deep vein thrombosis.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Each patient included to the study will undergo Point-of-Care ultrasound testing specific for the area defined in the Groups section.

SUMMARY:
The purpose of this study is to evaluate reliability of Point-of-Care ultrasound evaluation performed by general practitioners.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate reliability of Point-of-Care ultrasound (POCUS) evaluation performed by general practitioners.

General practitioners who underwent predefined training in POCUS will perform ultrasound examination in outpatients meeting inclusion criteria. While this is observational study, result will not have an impact on the management of the patients.

Regardless of the POCUS examination, patients undergo a routine diagnostic process which is appropriate for the initial symptom. Imaging examinations will always be a part of this. This will serve as an expert control to evaluate the reliability of POCUS Each POCUS examination will also be recorded as a video loop, subsequently assessed by an expert in the POCUS and also used as an expert control.

The data will be analyzed by standard reliability testing.

ELIGIBILITY:
Inclusion Criteria:

* Patient with abdominal pain in the right upper quadrant (will be indicated for the abdominal ultrasound) or patient with dyspnoea (will be indicated for lung ultrasound) or patient with suspected deep vein thrombosis (will be indicated for compression ultrasound testing)
* Signing of informed consent to participate in the study

Exclusion Criteria:

* Age <18 years
* Refusal of ultrasound examination by patient
* Any circumstance that prevents ultrasonographic examination (eg allergy to ultrasonographic gel, skin lesions that do not allow safe examination, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult outpatients.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Reliability of Point-of-Care ultrasound investigation of the lungs, gall bladder or proximal deep veins of lower extremities performed by general practitioner compared with the expert diagnostic method | 7 months
  General practitioners will perform the type of Point-of-Care ultrasound investigation which will relate to the type of symptoms. Then, the result of this investigation will be compared with the expert diagnostic method. This will be chest X ray scan or pulmonary CT for group 1 patients, expert abdominal ultrasound for group 2 patients and expert complete compression ultrasound for group 3 patients. These examinations are not study interventions, while they are a routine procedures, which would be indicated irrespective of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Skulec, MD, PhD, Principal Investigator — Masaryk Hospital Usti nad Labem
Locations (1):
- Masaryk Hospital Usti nad Labem, Ústí nad Labem, Czechia

REFERENCES:
- [Derived] Halata D, Zhor D, Skulec R, Seifert B. Accuracy of point-of-care ultrasound examination of the lung in primary care performed by general practitioners: a cross-sectional study. BMC Prim Care. 2025 Apr 8;26(1):99. doi: 10.1186/s12875-025-02802-4. PMID 40200132